CLINICAL TRIAL: NCT02154464
Title: Morphine-sparing Effect of Intravenous Paracetamol for Post-operative Pain Management Following Laparoscopic Gastric Banding in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Zlotnik, Professor, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR 0024-14 CTIL
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Morphine-sparing; Paracetamol; Obesity; Gastric banding
MeSH Terms: conditions — Obesity | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators predict that giving patients paracetamol in the operative period will reduce their need for opioid pain reducers in the post operative setting.

DETAILED DESCRIPTION:
This study is designed as a population-based prospective, double blind cohort study. A prospective cohort of patients admitted to laparoscopic gastric banding due to morbid obesity

STUDY GOALS

* To evaluate the morphine-sparing effect of paracetamol IV in obese patients undergoing bariatric surgery.
* To identify potential ability of paracetamol IV to attenuate or relief postoperative pain in obesity patient undergoing bariatric surgery
* To determine effectiveness of paracetamol IV to reduce postoperative complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients admitted for laparoscopic gastric banding
* Elective surgery
* BMI > 40
* ASA (American Society Anesthesiologists perioperative risk stratification) class 1-2

Exclusion Criteria:

* Patients' refusal to participate in the study
* Patients unable to give an informed consent
* Pregnancy
* Emergent surgery
* Patient with known allergy to morphine or paracetamol
* Patient with hepatic failure (based on history or elevated liver enzymes).
* ASA class >2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
amount of morphine | Until discharge (participants will be followed for the duration of hospital stay, an expected average of 3 days)
  The primary outcome will be the comparison amount of morphine injected in each group until discharge

SECONDARY OUTCOMES:
Complication during treatment of patient in PACU: | Until discarge from PACU (participants will be followed for the duration of PACU stay, an expected average of 2 hours)
  Complication during treatment of patient in PACU, including:
  * Respiratory complications (respiratory support, need for ICU, etc)
  * Cardiovascular complications (hemodynamic instability, inotropic support )
  * Gastrointestinal complications (nausea and vomiting tested by PONV scale, need to use antiemetic drugs)
  * Incidence of urinary retention and need for catheterization
  * Pruritus
Time discharging from PACU | Until discharge from PACU (participants will be followed for the duration of PACU stay, an expected average of 2 hours)
Length of hospitalization | Until discharge from hospital (participants will be followed for the duration of hospital stay, an expected average of 3 days)
Complications during hospitalization. | Until discharge from hospital (participants will be followed for the duration of hospital stay, an expected average of 3 days)
  Complications during hospitalization, including :
  * Septic complications
  * Respiratory, cardiac or other complications

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Ben Gurion University of the Negev, Beersheba, Israel

REFERENCES:
- [Derived] Semyonov M, Bartulovic A, Cohen N, Berzon B, Fedorina E, Lerman S, Semionov A, Friger M, Acker A, Geftler A, Zlotnik A, Brotfain E. The effect of timing of intravenous paracetamol on perioperative pain and cytokine levels following laparoscopic bariatric surgery, a randomized controlled trial. Obesity (Silver Spring). 2022 Nov;30(11):2185-2193. doi: 10.1002/oby.23545. Epub 2022 Sep 25. PMID 36161276